CLINICAL TRIAL: NCT00259597
Title: Morphometry of Breast Cells in Ductal Lavage
Brief Title: Nuclear Morphology of Breast Cells in Ductal Lavage
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Principal Investigator, Zora Djuric, Research Professor, University of Michigan
Other Study IDs: Morphology; 1R21CA100575-01A1 (NIH)
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2008-11

CONDITIONS: Benign Breast Disease
Keywords: nuclear morphology; image analysis; lipid peroxidation; diet; proliferative breast disease
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: breast ductal lavage — breast ductal lavage and nipple aspiration done once

SUMMARY:
Breast nipple aspirate fluids (NAF) are useful for non-invasive monitoring of the breast. NAF has been shown to exhibit large inter-individual differences in lipid peroxidation. Unfortunately, the yield of epithelial cells in NAF is low. More recently, breast ductal lavage has been approved for clinical use. Nuclear morphologic features of breast biopsies have been shown previously to have prognostic value for breast cancer risk. In women without cancer, there may be subtle changes in the breast epithelial cells that can only be defined with computer-assisted measurements. The subjects selected for this study will be 98 women with biopsy-confirmed proliferative breast disease. These women are at slightly increased breast cancer risk, and exhibit higher mean levels of cholesterol and cholesterol oxides in NAF than women with non-proliferative histology in the breast. Levels of 8-isoprostane, cholesterol, fatty acids, fat-soluble micronutrients and 2,6-cyclolycopene-4,5-diol will be quantified in breast NAF that is obtained before breast lavage. These measures were chosen based on their potential relationship to dietary intakes and to oxidative stress, which is relevant to the application of these methods to dietary prevention studies.The investigators will characterize the morphology of breast epithelial cells from lavage using quantitative image cytometry to capture nuclear and cellular area, diameter, roundness, perimeter, and nuclear:cytoplasmic area ratio. Correlations will be evaluated between the measured morphologic features and each analyte in the NAF. The impact of various clinical, demographic and dietary factors on cellular morphology will also be explored. This study will help establish the feasibility of using these measures as endpoints in dietary intervention studies and will generate hypotheses that should be tested in larger studies. Such measures also should be applicable to molecular epidemiological investigations that seek to examine the impact of certain gene polymorphisms and environmental exposures on biomarkers of cancer risk.

DETAILED DESCRIPTION:
WHY THE STUDY IS BEING DONE

Breast nipple aspirate fluids (NAF) can be obtained non-invasively from women, making analyses of this fluid relevant to studies of breast cancer risk. The inter-individual variation for lipid oxidation products (a type of damage to fats) in NAF is more than 100-fold, and these oxidation products are likely to have a toxic effect on the breast epithelial cells. During breast ductal lavage, NAF is first aspirated, and the ducts producing fluid are then subjected to lavage to obtain epithelial cells. The nuclear features (morphology) of these cells can then be examined. Nuclear morphology is a quantitative method to observe subtle changes in nuclear features, and these measures in benign breast biopsies have been shown to have prognostic value for breast cancer risk.

This exploratory study will help establish the feasibility of using these measures as endpoints in dietary intervention studies. Since the differences in lipid oxidation levels in NAF are markedly large, it is reasonable to believe that there must be some influence on nuclear morphology. These measures also should be applicable to investigations that seek to examine the impact of certain genetic polymorphisms and environmental exposures on biomarkers of oxidative stress and breast cancer risk.

We will study women who have been diagnosed previously with proliferative breast disease. These women may be good candidates for dietary prevention studies since they are at somewhat increased risk of breast cancer, receive little beyond surgery for treatment, and have been shown to have higher levels of lipid oxidation in the breast than women with no such diagnosis.

WHAT WE HOPE TO ACCOMPLISH

We hope to determine the feasibility of obtaining and analyzing both NAF and breast epithelial cells from women with benign proliferative breast disease. These women are at increased breast cancer risk, and the composition of the NAF, which bathes the breast ducts may affect the morphological features of the nuclei in the breast epithelial cells. If the levels of lipid oxidation products are higher in women with large nuclei (a risk factor for breast cancer), then interventions which reduce oxidative stress and cancer risk may be planned in the future.

The aims are:

1. To determine if levels of fats, damaged or oxidized fats, oxidized or damaged vitamins and vitamins (8-isoprostane, cholesterol, fatty acids, tocopherols, carotenoids and 2,6-cyclolycopene-4,5-diol) can be quantified in breast NAF obtained before breast lavage. Levels in NAF will be compared to that in blood. These measures were chosen based on their potential relationships to dietary intakes and to oxidative stress levels, which is relevant to intervention studies. Tocopherols and carotenoids are dietary antioxidants, and certain fatty acids are oxidized more readily than others. Both 8-isoprostane and 2,6-cyclolycopene-4,5-diol appear to be markers of oxidative stress.
2. To obtain breast lavage fluids from women with proliferative breast disease and to characterize the nuclear morphology of breast epithelial cells in the breast lavage fluid. We will quantify various measures commonly used in biopsies including nuclear diameter, circumference, area, roundness and nuclear:cytoplasmic area ratio. These measures have been shown to be related to breast cancer risk. If there are sufficient cells, analysis of oxidative DNA damage will be made using the comet assay.
3. To examine whether nuclear morphology is associated with levels of oxidative stress in the NAF. Correlations will be evaluated with levels of 8-isoprostane, cholesterol, specific fatty acids, 2,6-cyclolycopene-1,5-diol and fat-soluble micronutrients. The potential influence of diet, demographic factors and nature of previous biopsy diagnosis on nuclear morphology will also be examined as a sub-aim in an effort to better understand differences among women in the nuclear morphology of epithelial cells from ductal lavage.

The materials gathered for research purposes will be:

Consent Form Health Status Questionnaire Food Frequency Questionnaire Height and body weight Breast nipple aspirate fluid Breast lavage fluid 10-ml Blood sample biopsy date, diagnosis and history of medical problems from the medical chart

SAMPLE SIZE

It was desired to equip our study so that the variables of interest can be determined within a coefficient of variation (CV) of 25%, with 90% confidence. Sixty subjects would yield estimates of the mean level of 8 of the 9 study variables to within a CV of 25%, with 90% confidence. The one exception is the highly variable 8-isoprostane measure, whose mean level could be estimated to within a CV of 37%, with 90% confidence.

HOW THE STUDY WILL BE CONDUCTED

A total of 75 women will be recruited for this study over roughly 13 months (ten months of year 1 and 3 months of year 2) by a clinician. She will confirm from the patient chart the previous diagnosis of proliferative breast disease, obtain the type of breast disease diagnosed, how long ago it was diagnosed to the nearest month, and any breast or health problems that could affect the lavage results. The study subjects will fill out questionnaires, be weighed and measured for height, donate a 10-ml blood sample and undergo a breast lavage procedure. During the lavage procedure, breast nipple fluid and the lavage fluid will be collected.

Breast ductal lavage is an important new procedure that can be used to help determine a woman's risk for breast cancer. It is an attractive diagnostic method since it is associated with very little discomfort. At present, it is only used in certain women who are thought to be at very high-risk for breast cancer. During the ductal lavage procedure, the fluid-producing ducts must first be identified. This is done by first freeing the ducts at the nipple surface of keratin plugs, and a woman then uses massage to produce fluid. This fluid, called nipple aspirate fluid (NAF), is what bathes the breast ducts and will be collected for analysis in this proposed project. Once the ducts that produce NAF are identified, the physician then lavages the duct. The lavage fluid washes out breast cells that can then be evaluated by a pathologist to determine whether or not they are normal. The entire procedure is done using anesthetic at the nipple surface initially and in the lavage fluid to minimize any discomfort, and levels of discomfort is generally less than that with a mammogram.

An early indicator of breast cancer risk may be the characteristics of the epithelial cells from the lavage fluid. These breast cells are dislodged upon lavage, they are placed onto a slide and a pathologist examines them for abnormalities. Beyond the pathological diagnosis, there may be subtle changes in the appearance of the cells. Changes in the size and shape of the cell nucleus can be measured using a computer-driven microscope that has quantitative image analysis software. Increases in nuclear area, diameter and perimeter and less uniform roundness of nuclei are known to be associated with breast cancers of higher grade. These kinds of measures have also been measured in breast biopsies that were either normal or hyperplastic, and those women with larger nuclei in completely benign breast biopsies were more likely to develop breast cancer 1-33 years later.

One factor that may affect the shape of nuclei in breast cells is the level of oxidative stress in the breast. The breast fluid is very rich in fats, or lipids, and certain kinds of lipids are easily oxidized. NAF also contains vitamins obtained from fruits and vegetables that function as antioxidants to stop lipid oxidation. For example, carotenoids can react with harmful oxidants to form oxidized carotenoids. We will therefore measure levels of one lipid peroxidation marker and one oxidized carotenoid in NAF as markers of oxidative stress. We also will measure fatty acid levels and levels of un-oxidized carotenoids. We then will determine if differences in the composition of the NAF are related to the measures of nuclear shape made on breast cells.

The breast NAF and blood will be analyzed for cholesterol using spectrophotometric kits. Fatty acids will be analyzed using gas chromatography. Total 8-isoprostanes will be analyzed by immunoassay kits. Micronutrients and vitamins will be analyzed by high pressure liquid chromatography. Nuclear morphology will be analyzed by a computer-driven microscope. DNA damage in breast cells will be analyzed using gel electrophoresis of lysed cells (comet assay). Statistical analyses will allow us to determine if the NAF and blood measures are related to each other and to the nuclear measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* A diagnosis of proliferative breast disease
* At least 1 month post biopsy
* At least 3 months post any therapy such as tamoxifen
* Good general health
* Sign Consent Form.

Exclusion Criteria:

* Pregnant or lactating (lactation must have stopped at least 3 months prior)
* Taking coumadin
* Any diseases including cardiovascular, high blood pressure and diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women with a previous biopsy of proliferative breast disease
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zora Djuric, PhD, Principal Investigator — University of Michigan
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Result] Djuric Z, Edwards A, Madan S, Darga L, Ren J, Blake C, Koletsky M, Heilbrun LK. Obesity is associated with atypia in breast ductal lavage of women with proliferative breast disease. Cancer Epidemiol. 2009 Oct;33(3-4):242-8. doi: 10.1016/j.canep.2009.07.003. Epub 2009 Jul 28. PMID 19683484